CLINICAL TRIAL: NCT00108186
Title: Celecoxib-Mediated Inhibition of T Regulatory Cells in Human Lung Cancer
Brief Title: Celecoxib Treatment for Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Couldn't accrue patients
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other); City of Hope Medical Center (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONCA-043-04S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: cyclooxygenase 2; lung cancer; lymphocytes; non small cell; therapeutics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Other): Celecoxib is an FDA approved drug for other indications such as osteoarthritis. It is not FDA approved for non-small cell lung cancer.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — Eight subjects will be assigned to one of three cohorts. Subjects will receive Celecoxib in escalating doses per cohort, starting with 200mg twice a day by mouth; 400mg twice a day by mouth; and increasing to 600mg twice a day by mouth, for a total of 7 days. Subjects will have blood taken before the start of Celecoxib, and after completion of 7-days of Celecoxib.

SUMMARY:
This proposal evaluates cyclooxygenase 2 (COX-2) inhibition as a means to decrease T regulatory cell activities and thus augment immune responses against lung cancer. The broad goal focuses on understanding how COX-2 expression regulates the malignant phenotype in non small cell lung cancer in an effort to foster an informed approach for the use of COX-2 inhibitors in prevention and therapy for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed and surgically resectable non small cell lung cancer and subjects must be ineligible for or refuse, neoadjuvant therapy

Exclusion Criteria:

Hypersensitivity to celecoxib or NSAIDs, previous history of GI bleeding or ulceration, chronic or concurrent use of steroids and renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Measure bio-markers; safety measures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Dubinett, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States